CLINICAL TRIAL: NCT01586923
Title: A Prospective Study of RBC Transfusion in Children With Severe Anemia
Brief Title: RBC Transfusion in Severe Anemia With Lactic Acidosis
Acronym: TOTAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Walter H. Dzik, Co-Director, Blood Transfusion Service, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Anemia
Keywords: Anemia; Transfusion; RBC storage age; Tissue oxygenation; Malaria
MeSH Terms: conditions — Anemia; Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short-storage RBC (Active Comparator): RBC transfusion using packed RBCs stored for 10 days or less.
  Interventions: Biological: RBC transfusion
- Prolonged-storage RBC (Active Comparator): RBC transfusion using packed RBCs stored for 25 days or more.
  Interventions: Biological: RBC transfusion

INTERVENTIONS:
Biological: RBC transfusion — RBC transfusion of different storage age

SUMMARY:
The hypothesis of this study is that prolonged-storage RBCs are not inferior to short-storage RBCs for the time required to clear elevated blood lactate levels in children with severe anemia.

DETAILED DESCRIPTION:
This study will measure the time to resolution of lactic acidosis in patients with severe anemia following blood transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 mos to 5 years
* Hg < 5 g/dL and Lactate > 5 mM

Exclusion Criteria:

* Receiving transfusion other than RBCs
* Children with known or suspected cardiac disease

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 290 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Reduction of elevated levels of blood lactate during 24 following RBC transfusion | 24 hours

SECONDARY OUTCOMES:
Normalization of vital signs | 24 hours
Correction of acidosis | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Walter H Dzik, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mulago Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No
Data published

REFERENCES:
- [Derived] Dhabangi A, Ainomugisha B, Cserti-Gazdewich C, Ddungu H, Kyeyune D, Musisi E, Opoka R, Stowell CP, Dzik WH. Effect of Transfusion of Red Blood Cells With Longer vs Shorter Storage Duration on Elevated Blood Lactate Levels in Children With Severe Anemia: The TOTAL Randomized Clinical Trial. JAMA. 2015 Dec 15;314(23):2514-23. doi: 10.1001/jama.2015.13977. PMID 26637812